CLINICAL TRIAL: NCT05339659
Title: Design and Testing of a mHealth App for Ambivalent Smokers Living With HIV: A Randomized Pilot Study
Brief Title: Randomized Pilot Study of a mHealth App for Ambivalent Smokers Living With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Jennifer McClure, Director of Research, Faculty & Development, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: R21CA261199 (NIH)
Record Dates: First submitted 2022-04-11; First posted 2022-04-21 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Smoking; Smoking Cessation
Keywords: HIV
MeSH Terms: conditions — Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): mHealth app consisting of standard, best-practice information and guidance to help people stop smoking.
  Interventions: Device: mHealth Intervention
- Experimental (Experimental): mHealth app consisting of standard, best-practice information and guidance to help people stop smoking + additional experimental content targeted to smokers living with HIV who are ambivalent about quitting smoking.
  Interventions: Device: mHealth Intervention

INTERVENTIONS:
Device: mHealth Intervention — Mobile health (mHealth) app to motivate and support quitting smoking.

SUMMARY:
This pilot study will assess the acceptability and feasibility a novel mHealth app designed for smokers who are ambivalent about quitting and have been diagnosed with HIV.

DETAILED DESCRIPTION:
This study will use a randomized, parallel, two-arm trial to compare outcomes between people assigned to use a "standard care" mHealth app versus a similar app with additional content targeted to people living with HIV. A total of up to 50 people will be enrolled and followed for three months to assess outcomes.

ELIGIBILITY:
Inclusion Criteria Include:

* 18 years of age or older;
* Comfortable speaking and reading in English;
* Smoked at least 100 cigarettes in their lifetime;
* Smoked, even a puff, in the past 7 days;
* Smoked at least 5 cigarettes a day;
* Are interested in quitting smoking someday, but not in the next month;
* Have an iPhone Operating System (iOS) or Android smart phone which they use at least weekly;
* Are willing to upgrade their phone operating system, if needed;
* Agree to download and try the app;
* Do not use Virtual Private Network (VPN) on their smart phone;
* Live in the United States and have a valid U.S.-based mailing address and phone number;
* Have been diagnosed with HIV

Exclusion Criteria Include:

* Refusing to answer all screening questions
* History of dementia or psychosis
* Visual impairments that preclude their ability to view content on their smart phone and lack adaptive devices to view content
* Contraindications for nicotine replacement therapy (NRT) use (e.g., based on medical history or daily smoking level)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McClure, PhD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente WA Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McClure JB, Heffner JL, Krakauer C, Mun S, Catz SL. A Novel mHealth App for Smokers Living With HIV Who Are Ambivalent About Quitting Smoking: Formative Research and Randomized Feasibility Study. JMIR Form Res. 2024 Jul 8;8:e58063. doi: 10.2196/58063. PMID 38976321

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment began 06/02/2022 and study activities completed 05/20/2023. Participants were recruited through: (1) social media advertisements; (2) direct outreach to Kaiser Permanente Washington members living with HIV; (3) ResearchMatch.org; (4) partnership with various HIV/AIDS service organizations; and (5) community health clinics in the Seattle area.
Pre-assignment Details: Twenty-two participants were consented and randomized, of whom 19 ultimately installed the study app and were thus eligible for inclusion in the analytic cohort. Because app installation is a metric of feasibility, we report on both on the number who enrolled (N=22) and were used to assess app installations and the number in the final analytic cohort (N=19).
Period: Overall Study
Arm/Group | Control | Experimental
Started | 9 (Number in control arm screened as eligible and randomized.) | 13 (Number in experimental arm screened as eligible and randomized.)
Installed App | 7 (Number who installed the app and was included in the analytic cohort for outcome analyses.) | 12 (Number who installed the app and were included in the analytic cohort for the outcome analyses.)
Completed 1-month Self-report Survey | 6 | 9
Completed 3-month Self-report Survey | 6 | 8
Completed App Utilization Period | 7 | 12 (Twelve participants completed the app utilization period. However, complete app utilization data was only available on 11 participants; one participant had incomplete data due to a technical issue.)
Completed | 7 | 12
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Experimental | Total
Number analyzed (Participants) | 7 | 12 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (10.7) | 49.6 (12.5) | 49.3 (11.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female gender | 0 | 2 | 2
  Male gender | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 12 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 6 | 7 | 13
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes/day] | 10.3 (3.5) | 11.9 (5.2) | 11.3 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Intervention (App) Utilization
Description: Number of unique app user-sessions
Time Frame: 3 months post-enrollment
Population: All individuals who installed the app and were not administratively removed (n=19).
Measure: Mean (Standard Deviation); unit: User sessions
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 12
User sessions | 4.9 (1.3) | 8.2 (6.9)
Statistical Analysis 1: Comparison: Control vs Experimental; A priori power calculations estimated detectable differences with 80% power with type 1 error rate=0.05, assuming a two-sided unequal variance t-test (standard deviations of 2.0 and 7.0 in the control and experimental arms, respectively) and a total sample of n=50 equally split between arms. Given a final sample size of 19 (7 control, 12 experimental), we re-calculated the detectable mean difference with these sample sizes (maintaining all other original assumptions), which is 6.51 sessions; Test type: Other — The point null hypothesis of the significance test was a difference in expected number of log ins of 0; p = 0.219, Regression, Linear; Mean Difference (Final Values) = 3.55, 95% CI 2-sided [-2.33 to 9.44] — mean difference=experimental-control

2. Secondary Outcome: App Installation and Use
Description: Number of people in each study arm who installed the assigned app and used it at least one time. These people were included in the analytic cohort used to analyze all other study outcomes.
Time Frame: 3 month follow-up
Population: Individuals randomized to either arm who were not administratively removed (n=22).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 9 | 13
Participants | 7 | 12

3. Secondary Outcome: App Utilization - Cumulative Days of Use
Description: Cumulative number of days between the first and last use of the assigned app
Time Frame: 3 month follow-up
Population: All individuals who installed the app and were not administratively removed (n=19).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 12
days | 54.3 (39.8) | 30.4 (20.6)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in average number of days of use between arms; p = 0.153, Regression, Linear; Mean Difference (Final Values) = -22.12, 95% CI 2-sided [-53.44 to 9.19] — mean difference=experimental-control

4. Secondary Outcome: Self-reported 24-hour Quit Attempt
Description: At least one intentional smoking quit attempt lasting at least 24 hours. Missing outcomes imputed as not making a quit attempt.
Time Frame: 3 months post-enrollment
Population: Individuals who installed the app and were not administratively removed (n=19).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 12
Participants | 4 | 8
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is a relative difference=0; p = 0.727, Barnard's exact test; Risk Difference (RD) = 0.095, 95% CI 2-sided [-0.352 to 0.558] — risk difference=experimental-control

5. Secondary Outcome: Satisfaction With App Content and Advice
Description: Satisfaction with the overall "content and advice" of the assigned app, rated on a Likert scale from 1="not at all satisfied" to 5="extremely satisfied".
Time Frame: 1 month follow-up
Population: Participants who installed the app, were not administratively removed, responded to the question in the 1-month survey, and earned at least 1 badge by the time of the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 3 | 8
score on a scale | 3.0 (0.0) | 3.5 (0.8)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in average score between arms; p = 0.325, Regression, Linear; Mean Difference (Final Values) = 0.50, 95% CI 2-sided [-0.60 to 1.61] — mean difference=experimental-control

6. Secondary Outcome: Satisfaction With App Content and Advice
Description: as for outcome 5
Time Frame: 3 month follow-up
Population: Participants who installed the app, were not administratively removed, responded to the question in the 3-month survey, and earned at least 1 badge by the time of the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 4 | 7
score on a scale | 3.2 (1.3) | 3.6 (0.8)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis of the significance test is 0 difference in average score between arms; p = 0.745, Regression, Linear; Mean Difference (Final Values) = 0.22, 95% CI 2-sided [-1.28 to 1.72] — mean difference=experimental-control

7. Secondary Outcome: Earned Nicotine Replacement Therapy (NRT)
Description: Positive indicator if participants earn minimum number of badges required to receive free nicotine replacement therapy
Time Frame: 3 month follow-up
Population: 19 (7 control and 12 experimental) participants installed the app and were not administratively removed.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 12
Participants | 0 | 7
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis of the significance test is a risk difference=0; p = 0.009, Barnard's exact test; Risk Difference (RD) = 0.58, 95% CI 2-sided [0.16 to 0.85] — risk difference=experimental-control

8. Secondary Outcome: Not Smoking (Even a Puff) in the Last 7 Days
Description: 7-day point prevalent abstinence: self-report of not smoking, even a puff, in the last 7 days. Missing values were imputed as smoking.
Time Frame: 3-months post-enrollment
Population: All individuals who installed the app and were not administratively removed (n=19).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 12
Participants | 0 | 0

9. Secondary Outcome: Proportion Who Request Nicotine Replacement Therapy
Description: Among participants eligible to receive free nicotine replacement therapy based on their app use, how many request it in each study arm.
Time Frame: 3 month follow-up
Population: Participants who received enough badges to earn free NRT; no participants in the control arm met these criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 0 | 7
Participants | 0 | 0

10. Secondary Outcome: Number of Cigarettes Smoked Per Day
Description: Self-reported average number of cigarettes smoked per day at follow-up
Time Frame: 1 month follow-up
Population: Participants who installed the app, were not administratively removed, and responded to the question in the 1-month survey.
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | Control | Experimental
Number analyzed (Participants) | 6 | 9
cigarettes/day | 7.2 (3.4) | 8.6 (6.7)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is a mean difference of 0 cigarettes/day between arms; p = 0.469, Regression, Linear; Adjusted for baseline cigarettes/day; Mean Difference (Final Values) = 1.39, 95% CI 2-sided [-2.66 to 5.44] — mean difference=experimental-control

11. Secondary Outcome: Number of Cigarettes Smoked Per Day
Description: Self-reported average number of cigarettes smoked per day at follow-up
Time Frame: 3 month follow-up
Population: Participants who installed the app, were not administratively removed, and responded to the question in the 3-month survey.
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | Control | Experimental
Number analyzed (Participants) | 5 | 8
cigarettes/day | 7.4 (3.4) | 7.9 (3.6)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is a mean difference of 0 cigarettes/day between arms; p = 0.614, Regression, Linear; Adjusted for baseline cigarettes/day; Mean Difference (Final Values) = -0.66, 95% CI 2-sided [-3.48 to 2.16] — mean difference=experimental-control

12. Secondary Outcome: Motivation for Quitting Smoking
Description: Self-reported motivation for quitting smoking or remaining quit assessed using a 10 point Likert scale from 1=not at all to 10=extremely.
Time Frame: 1 month follow-up
Population: Participants who installed the app, were not administratively removed, and responded to the question about motivation for quitting in the 1-month survey (n=15).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 6 | 9
score on a scale | 7.5 (2.5) | 6.8 (2.7)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in average score between arms; p = 0.90, Regression, Linear; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-2.67 to 2.38] — mean difference=experimental-control

13. Secondary Outcome: Motivation for Quitting Smoking
Description: as for outcome 12
Time Frame: 3 month follow-up
Population: Participants who installed the app, were not administratively removed, and responded to the question about motivation to quit in the 3-month survey (n=14).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 6 | 8
score on a scale | 7.8 (1.9) | 6.8 (1.8)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in average score between arms; p = 0.632, Regression, Linear; Mean Difference (Final Values) = -0.55, 95% CI 2-sided [-3.03 to 1.93] — mean difference=experimental-control

14. Secondary Outcome: Self-efficacy for Quitting Smoking
Description: Self-reported confidence in one's ability to quit smoking assessed using a 10 point Likert scale item ranging from 1=not at all to 10=extremely.
Time Frame: 1 month follow-up
Population: Participants who installed the app, were not administratively removed, and responded to the question in the 1-month survey about self-efficacy to quit smoking (n=15).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 6 | 9
score on a scale | 8.3 (2.1) | 6.2 (1.5)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in average score between arms; p = 0.227, Regression, Linear; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-3.55 to -0.94] — mean difference=experimental-control

15. Secondary Outcome: Self-efficacy for Quitting Smoking
Description: as for outcome 14
Time Frame: 3 month follow-up
Population: Participants who installed the app, were not administratively removed, and responded to the question about self-efficacy to quit smoking in the 3-month survey (n=13).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Experimental
Number analyzed (Participants) | 5 | 8
score on a scale | 8.6 (1.5) | 7.0 (1.8)
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in average score between arms; p = 0.274, Regression, Linear; Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-3.58 to 1.15] — mean difference=experimental-control

16. Other Pre Specified Outcome: Utilization - Personal Experiments
Description: Number of "personal experiment" exercises completed in the experimental arm out of a maximum of 10.
Time Frame: 3 month follow-up
Population: Participants in the experimental arm who installed the app and were not administratively removed (n=12).
Measure: Mean (Standard Deviation); unit: experiments
Arm/Group | Experimental
Number analyzed (Participants) | 12
experiments | 3.7 (3.3)

17. Other Pre Specified Outcome: Quit Guide Participation
Description: Earning at least one badge from the quit guide (one possible with each of 6 steps to the quit guide).
Time Frame: 3 month follow-up
Population: Participants who installed the app, were not administratively removed, and whose data we were able to track (technical issues removed one individual for this reason from the experimental arm).
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 11
Participants | 4 | 1

18. Other Pre Specified Outcome: Quit Guide Completion
Description: Earning all 6 badges possible from the quit guide (one badge earned for each of 6 total steps completed).
Time Frame: 3 month follow-up
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 11
Participants | 0 | 0

19. Other Pre Specified Outcome: Cigarette Tracker Use
Description: Use of the cigarette tracker tool (earning the badge for use).
Time Frame: 3 month follow-up
Population: Participants who installed the app and were not administratively withdrawn.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 12
Participants | 1 | 3
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in probability of engaging with the app component; p = 0.981, Barnard's exact test; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.39 to 0.39] — risk difference=experimental-control

20. Other Pre Specified Outcome: Savings Calculator Use
Description: Use of the savings calculator tool (earning the badge for use).
Time Frame: 3 month follow-up
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 11
Participants | 2 | 3
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in probability of engaging with the app component; p = 0.845, Barnard's exact test; Risk Difference (RD) = -0.01, 95% CI 2-sided [-0.49 to 0.43] — risk difference=experimental-control

21. Other Pre Specified Outcome: Read Peer Testimonials
Description: Indication that each provided peer testimonial on how to talk back to common excuses for not quitting was opened and viewed.
Time Frame: 3 month follow-up
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 11
Participants | 1 | 1
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in probability of engaging with the app component; p = 0.560, Barnard's exact test; Risk Difference (RD) = -0.05, 95% CI 2-sided [-0.47 to 0.28]; risk difference=experimental-control

22. Other Pre Specified Outcome: Read Peer Advice
Description: Indication that each page of the peer advice and motivational support vignette was opened and viewed.
Time Frame: 3 month follow-up
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 11
Participants | 1 | 2
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in probability of engaging with the app component; p = 0.981, Barnard's exact test; Risk Difference (RD) = 0.04, 95% CI 2-sided [-0.39 to 0.39] — risk difference=experimental-control

23. Other Pre Specified Outcome: Journal Opened
Description: Indication the journal was opened at least one time.
Time Frame: 3 month follow-up
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 11
Participants | 6 | 8
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in probability of engaging with the app component; p = 0.632, Barnard's exact test; Risk Difference (RD) = -0.13, 95% CI 2-sided [-0.49 to 0.34] — risk difference=experimental-control

24. Other Pre Specified Outcome: Use of More Help Feature
Description: Indication the More Help page (with contact information for a tobacco quit-line and more resources for quitting smoking) was viewed at least one time
Time Frame: 3 month follow-up
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Experimental
Number analyzed (Participants) | 7 | 11
Participants | 4 | 6
Statistical Analysis 1: Comparison: Control vs Experimental; Test type: Other — The null hypothesis for the significance test is 0 difference in probability of engaging with the app component; p > 0.999, Barnard's exact test; Risk Difference (RD) = -0.03, 95% CI 2-sided [-0.48 to 0.45] — risk difference=experimental-control

25. Other Pre Specified Outcome: Completing "Just the Facts" Toolbox Component
Description: Completing and earning the badge for the "just the facts" toolbox component; only available to the experimental arm.
Time Frame: 3 month follow-up
Population: Participants in the experimental arm who installed the app and were not administratively removed and whose data we were able to track (n=11).
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 11
Participants | 3

ADVERSE EVENTS:
Time Frame: For each participant, adverse events (AE's) were collected over a 3 month period, starting at baseline and ending at 3-month follow-up. Events were monitored continually during this period.
Arm/Group | Control | Experimental
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 0/7 | 0/12

LIMITATIONS AND CAVEATS:
The purpose of this pilot was to inform feasibility and acceptability of the experimental app among smokers who were ambivalent about quitting. Data were analyzed among participants who installed the app (n = 19) and are subject to missingness for some outcomes. This pilot study was not powered to provide definitive answers about the efficacy of the intervention. A larger trial is needed for this.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT05339659/Prot_SAP_000.pdf